CLINICAL TRIAL: NCT05948111
Title: Insights From Participants: Candid Accounts of Schizophrenia Clinical Trials Patients
Brief Title: Assessment of Schizophrenia Patients' Clinical Study Experiences
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 83338153
Record Dates: First submitted 2023-07-07; First posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Schizophrenia
Keywords: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study seeks to delve into the firsthand experiences of patients diagnosed with schizophrenia who partake in a separate clinical trial featuring a specific medical intervention. The primary emphasis will be on meticulously tracking the rates of trial completion and withdrawal among these individuals.

The data collected from this study will help improve future outcomes for all schizophrenia patients as well as those in under-represented demographic groups.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia
* Considered reliable, able to understand, and willing to perform all study procedures
* Signed Written Informed Consent

Exclusion Criteria:

* Currently enrolled in, have completed or have discontinued from a clinical trial involving an investigational drug
* Is pregnant, breastfeeding or expecting to conceive within the projected duration of the study
* Any serious and/or unstable pre-existing medical disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with schizophrenia who are actively considering enrolling in an observational clinical study for said condition, but have not yet completed enrollment and randomization phases.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Number of schizophrenia patients who decide to enroll in a clinical trial | 3 months
Rate of schizophrenia patients who remain in clinical trial to trial completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Runge K, Fiebich BL, Kuzior H, Saliba SW, Yousif NM, Meixensberger S, Nickel K, Denzel D, Schiele MA, Maier SJ, Berger B, Dersch R, Domschke K, Tebartz van Elst L, Endres D. An observational study investigating cytokine levels in the cerebrospinal fluid of patients with schizophrenia spectrum disorders. Schizophr Res. 2021 May;231:205-213. doi: 10.1016/j.schres.2021.03.022. Epub 2021 Apr 19. PMID 33887648
- [Background] Srisurapanont M, Kunchanaphongphan T, Chokemaitree N, Prachason T, Kanchanatawan B, Suttajit S, Sanguanvichaikul T, Trisukon W, Dendumrongkul P, Chinvararak C, Kawilapat S. Course and predictors of disability in Thai patients with schizophrenia: A 2-year, multi-center, prospective, observational study. Asian J Psychiatr. 2022 Apr;70:103044. doi: 10.1016/j.ajp.2022.103044. Epub 2022 Feb 19. PMID 35219052
- [Background] Garcia-Portilla MP, Benito Ruiz A, Gomez Robina F, Garcia Dorado M, Lopez Rengel PM. Impact on functionality of the paliperidone palmitate three-month formulation in patients with a recent diagnosis of schizophrenia: a real-world observational prospective study. Expert Opin Pharmacother. 2022 Apr;23(5):629-638. doi: 10.1080/14656566.2021.2023496. Epub 2022 Jan 5. PMID 34986711

DOCUMENTS (1):
  • Informed Consent Form (2023-07-07): https://cdn.clinicaltrials.gov/large-docs/11/NCT05948111/ICF_000.pdf